CLINICAL TRIAL: NCT02926391
Title: Evaluation of Safety and Efficency of Custom-made Corpectomy Implants: UNiD 3D VBR
Brief Title: UNiD 3D VBR Register
Status: Completed | Type: Observational
Sponsor: Medicrea International (Industry)
Responsible Party: Sponsor
Other Study IDs: 1801
Record Dates: First submitted 2016-06-27; First posted 2016-10-06 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Spinal Cord Compression; Spondylosis; Ossification of Posterior Longitudinal Ligament; Spinal Neoplasms; Bone Disease, Infectious
MeSH Terms: conditions — Spinal Cord Compression; Spondylosis; Ossification of Posterior Longitudinal Ligament; Spinal Neoplasms; Bone Diseases, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cervical: 30 patients who need anterior cervical corpectomy and fusion with patient-specific implants (UNiD 3D VBR)
  Interventions: Device: UNiD 3D VBR
- Thoraco-lumbar: 30 patients who need anterior thoracolumbar corpectomy and fusion with patient-specific implants (UNiD 3D VBR)
  Interventions: Device: UNiD 3D VBR

INTERVENTIONS:
Device: UNiD 3D VBR — Corpectomy of one or several vertebral body(ies) followed by vertebral body(ies) replacement and fusion
  Other Names: Patient-specific corpectomy implants; Custom-made corpectomy implants

SUMMARY:
Multicenter study allowing to include the first sixty patients implanted with a custom-made corpectomy implant (UNiD 3D VBR): 30 patient implanted in cervical region and 30 patients implanted in thoracolumbar region.

The main objective is to confirm feasibilty and safety of patient-specific implants for one or multi-level corpectomy and fusion.

This study was approved in March 2016 allowing to include retrospectivley all patients since the first implantation in January 2015 and prospectively all patients after the approval.

DETAILED DESCRIPTION:
Anterior cervical corpectomy with fusion (ACCF) has been demonstrated as a good alternative to anterior cervical discectomy and fusion (ACDF) to treat cervical spondylotic myelopathy (CSM). However, the use of vertebral body replacement (VBR) cages is technically demanding, especially to adjust the size of the cage to the defect without compromising the endplate integrity increasing the risk of subsidence. Beside recent studies advocating the interest of the shape, size and design of an implant to achieve fusion and stability in cervical spinal diseases indications, 3D printing offering rapid and patient-specific manufacturing has emerged over the past years. Several materials and technologies can be used and clinical and radiological data are still sparse.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent a single or multilevel cervical or thoracolumbar coprectomy and implanted with a patient specific implant (UNiD 3D VBR) for the following indications:

   * Cervical region

     * Fracture / Trauma
     * Tumors
     * Cervical spondylotic myelopathy
     * Infection (Ex: Osteomyelitis)
     * Spinal instability
     * Symptomatic degenerative spinal disease
     * Inflammatory rheumatism.
     * Pseudarthrosis
   * Thoracolumbar region

     * Fracture / Trauma
     * Tumors
     * Infection (Ex: Osteomyelitis)
     * Spinal instability
     * Symptomatic degenerative spinal disease
     * Pseudarthrosis
2. Patients > 18 years
3. Patients who signed an Informed Consent Form

Exclusion Criteria:

1. Patients who can't or doesn't want to sign an ICF
2. Patients unable to fill HRQOL questionnaires
3. Non-compliant paitents regarding follow-up or protocol
4. Pregnant patient or intended to be pregnant within the next 2 years
5. Sytemic or local infection
6. Allergy known or suspected to a componant
7. Patients presenting a contraindication as indicated in the instruction for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need single or multilevel corpectomy and fusion and who received a patient specific implants UNiD 3D VBR
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Quantification and description of implant-related adverse events | 12 months
  To confirm the safety of the surgery with patient specfic implant (UNiD 3D VBR). To quantify and describe adverse events or revision surgeries occuring during follow-up

SECONDARY OUTCOMES:
Fusion status | 6, 12, 24 months
  Radiological assessment of bony fusion
Length of surgery | During surgery
  Surgeon questionnaire will be used to quantify surgery's length
Surgical metrics | During surgery
  Surgeon questionnaire will be used to describe the surgery
Quality of life | preoperatively and 6,12, and 24 months postoperation
  mJOA: Modified Japanese Orthopaedic Association Score
Quality of life | preoperatively and 6,12, and 24 months postoperation
  EMS: European Myelopathy Score
Pain | preoperatively and 6,12, and 24 months postoperation
  Visual Analog Score
Disability | preoperatively and 6,12, and 24 months postoperation
  Neck disability index
Variation of radiological vertebral heights | 6,12, 24 months
  Xrays assessment of segmental height operated
Variation of radiological vertebral angulation | 6,12, 24 months postoperativley
  Xrays assessment of C2C7 angle and corpectomy angles

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Edouard Loret, MD, Principal Investigator — CHU Tours
Locations (1):
- CHU Tours, Tours, France

IPD SHARING:
Plan to Share IPD: No